CLINICAL TRIAL: NCT06952816
Title: Functional, Clinical, and Predictive Validation Study of the EMILY AI Device in Patients With Acute and Chronic Respiratory Failure
Brief Title: Validation Study of the EMILY AI Device in Acute and Chronic Respiratory Failure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aether Tech S.L. (Industry)
Collaborators: Hospital Universitario Fundación Jiménez Díaz (Other); Hospital Clinic of Barcelona (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FJD-EMILY-23-02
Record Dates: First submitted 2025-04-08; First posted 2025-05-01 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Chronic Respiratory Failure; Acute Respiratory Failure
Keywords: Respiratory failure; Hypoxia; Hyperxia; Oxigenotherapy
MeSH Terms: conditions — Respiratory Insufficiency; Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with respiratory failure (Experimental): Patients with respiratory failure who meet the inclusion criteria and none of the exclusion criteria.
  Interventions: Device: Emily.AI

INTERVENTIONS:
Device: Emily.AI — EMILY.AI is composed of an O2 regulating valve together with an intelligent system which allows the automation in the regulation of O2 and its customization.

SUMMARY:
Currently, there is no holistic solution for patients with respiratory diseases that includes oxygenation and management of a patient with respiratory disease, combining dynamic and automatic O2 administration and the detection of clinical worsening, generating a diagnostic suspicion, a management proposal, and notifying the medical team.

For device validation, prospective studies will be conducted in patients in respiratory intermediate care units, conventional hospitalization, during physical activity in the hospital setting, and in an out-of-hospital setting. The device will be evaluated in terms of oxygenation efficacy, response time, patient safety, efficiency, versatility, clinical benefit, and adaptability.

DETAILED DESCRIPTION:
There is no doubt about the efficacy of oxygen therapy in the treatment of acute and chronic respiratory failure in different clinical settings. However, its therapeutic dosage is not as strict as that of other treatments. Hypoxemia has been associated with increased mortality in multiple pathologies and clinical situations. Furthermore, the liberal use of oxygen therapy has also demonstrated harmful effects. Therefore, titration of this therapy is necessary. Traditionally, this has been performed manually, although in recent years, new devices have been developed to automatically adjust O2 flow rates to the needs of each patient, with the goal of maintaining stable oxygen saturations. These systems have the potential to reduce medical error, improve morbidity and mortality, and reduce care costs.

This study is a clinical investigation using a non-CE marked medical device, prospectively validating the device's functional status. The objective is to evaluate its efficacy and safety in patients with respiratory failure, both in hospital and outpatient settings.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 18 years of age.
* Admitted to intermediate respiratory care unit with a diagnosis of acute respiratory failure for at least 8 hours.
* Informed consent understood and signed.

Exclusion Criteria:

* Hemodynamic instability.
* Severe temperature changes.
* Hemoglobinopathies, severe anemia, severe acidosis, or severe alkalosis.
* Anatomical disturbances.
* Pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04-23 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
EFFICACY - EVALUATION OF THE RATE THE DEVICE MAINTAINS BLOOD OXYGEN SATURATION LEVELS | From enrollment to the end of treatment at 8 hours.
  Evaluation of the rate that the device maintains blood oxygen saturation levels measured by pulse oximetry within predetermined ranges in patients diagnosed with ARF (hypoxemic patients: 94-98%; hypercapnic patients: 92-94%) without providing less or more oxygen than required to keep the patient within the defined range.

SECONDARY OUTCOMES:
ACCURACY - MEASUREMENT OF THE SYSTEM'S ACTION SPEED CORRECTING THE OXYGEN SATURATION LEVELS | From enrollment to the end of treatment at 8 hours.
  Calculate the speed of action of the system from 1) detection of saturation out-of-range to the start of correction and 2) until the patient returns to the defined saturation range
ALERT SYSTEM - MEASUREMENT OF THE NUMBER OF SYSTEM ALERTS | From enrollment to the end of treatment at 8 hours.
  Measure the number of times EMILY alerts about a change in the oxygen saturation of monitored patients using its alarm system.
ALERT SYSTEM - EVALUATION OF THE AUTHENTICITY OF THE SYSTEM ALERTS BY COMPARING THE OXYGEN SATURATION LEVELS WITH A CONVENTIONAL SYSTEM | From enrollment to the end of treatment at 8 hours.
  Evaluate the alarm's authenticity by checking oxygen saturation with a conventional system and, in case of discrepancies, by arterial blood gas analysis.
EFFICIENCY - MEASUREMENT OF THE NUMBER OF TIMES THE MEDICAL AND NURSING TEAM MUST ADJUST THE OXYGENATION | From enrollment to the end of treatment at 8 hours.
  Evaluate the need for nursing and medical team intervention, measured by the number of times they must visit to adjust oxygenation or address symptoms related to oxygenation, primarily cardiorespiratory symptoms.
VERSATILITY - COMPARISON OF BLOOD OXYGEN SATURATION LEVELS MAINTENANCE BETWEEN DIFFERENT PROFILES AND SITUATIONS | From enrollment to the end of treatment at 8 hours.
  Evaluation of the rate that the device maintains blood oxygen saturation levels in different profiles, such as patients with pure hypoxemia and those with hypercapnia, and in different clinical situations such as bed rest, sitting, eating, or receiving physical therapy. This rate will be compared across these different profiles and situations.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Fundación Jiménez Díaz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided